CLINICAL TRIAL: NCT06444594
Title: Transient Receptor Potential Channels in Human Skin
Brief Title: Transient Receptor Potential Channels
Acronym: TRP
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Lacy Alexander, Professor of Kinesiology, Penn State University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 24921
Record Dates: First submitted 2024-05-24; First posted 2024-06-05 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Aging
MeSH Terms: interventions — Menthol; Camphor; Capsaicin; TRPV4 protein, human

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Vehicle Gel (Placebo Comparator): Non-active topical gel
  Interventions: Other: Vehicle gel
- Transient Receptor Potential (M8) Agonist (Experimental): Topical menthol gel applied once at 10%
  Interventions: Drug: TRPM8 Agonist
- Transient Receptor Potential (V4) Agonist (Experimental): Topical capsaicin gel applied once at 0.05%
  Interventions: Drug: TRPV4 Agonist
- Transient Receptor Potential (V1) Agonist (Experimental): Topical camphor gel applied once at 0.6%
  Interventions: Drug: TRPV1 Agonist
- Transient Receptor Potential M8 V4 V1 Agonist (Experimental): Topical menthol 10%, capsaicin 0.05%, camphor 0.6% applied once
  Interventions: Drug: TRPM8, TRPV4, TRPV1 Agonists
- no gel (No Intervention): no gel comparison

INTERVENTIONS:
Drug: TRPM8 Agonist — menthol gel 4-10%
  Other Names: menthol
  Arms: Transient Receptor Potential (M8) Agonist
Drug: TRPV1 Agonist — camphor gel 5-20%
  Other Names: camphor
  Arms: Transient Receptor Potential (V1) Agonist
Drug: TRPV4 Agonist — capsaicin gel 0.05-1%%
  Other Names: capsaicin
  Arms: Transient Receptor Potential (V4) Agonist
Drug: TRPM8, TRPV4, TRPV1 Agonists — menthol (4-10%), capsaicin (0.05-1%), camphor (5-20%)
  Other Names: menthol, capsaicin, camphor
  Arms: Transient Receptor Potential M8 V4 V1 Agonist
Other: Vehicle gel — Inactive vehicle gel
  Other Names: Inactive vehicle gel
  Arms: Vehicle Gel

SUMMARY:
Neurovascular signaling in the skin associated with stimulation of the transient receptor potential (TRP) channels. These channels are stimulated by both temperature and naturally occurring bioactive agents found in mint, chili peppers, garlic, etc. The aim of the study is to examine how topically applied TRP channel agonists including menthol, capsaicin and camphor impact neurovascular responses in the skin.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old.
* Women will not be pregnant and/or breastfeeding.

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Nicotine use (e.g., smoking, chewing tobacco etc.), quantified as more than 100 cigarettes or cigars in a lifetime)
* Known skin allergies or current rash, skin disease, disorders of pigmentation
* Diabetes
* Body mass index >35kg*m-2
* Using calcium channel blockers
* Raynaud's syndrome
* Allergy or hypersensitivity to menthol, camphor, capsaicin or adhesive
* Regular use (defined as greater than once a week) of topical analgesics that contain menthol, camphor or capsaicin

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin blood flow during slow local heating | 75 minutes
  Laser doppler flowmeter to measure skin blood flow during a slow local heating of the skin
Somatosensory perception | every 5 minutes for 120 minues
  heat and cold perception using a visual analog scale
algometer measurement | every 30 minutes for 120 minutes
  pain pressure thresholds

CONTACTS AND LOCATIONS:
Overall Officials: Lacy Alexander, Ph.D., Principal Investigator — Penn State University
Locations (1):
- Noll Laboratory, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No